CLINICAL TRIAL: NCT05989152
Title: Evolution of Positron Emission Computed Tomography (PET) Fixation With Fluorodeoxyglucose (FDG) at the End of Antibiotic Treatment of Infective Endocarditis on Valvular Prosthesis
Brief Title: Evolution of PET Fixation With FDG at the End of Antibiotic Treatment of Infective Endocarditis on Valvular Prosthesis
Acronym: EndEOTEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP230123; 2022-A02782-41 (Other: IDRCB)
Record Dates: First submitted 2023-05-24; First posted 2023-08-14 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Prosthetic Valve Endocarditis
Keywords: Infective endocarditis; end of treatment; Positron emission tomography
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Definite prosthetic valve endocarditis (Experimental): adult patients with a valvular prosthesis presenting a definite infective endocarditis (IE) according to the ESC classification in force, not operated on in the acute phase (before the PET scan at the end of treatment) and presenting a pathological FDG uptake on the prosthetic valve at the start of curative antibiotic treatment.
  Interventions: Radiation: FDG-PET at the end of treatment for IE

INTERVENTIONS:
Radiation: FDG-PET at the end of treatment for IE — FDG-PET at the end of treatment for IE in patients with a prosthetic valve

SUMMARY:
In patients with prosthetic valve endocarditis (PVE) and pathological valvular FDG uptake on the initial FDG-PET and not referred to valve replacement at the acute phase, the study will assess whether FDG-PET is able to identify those at increased risk of PVE relapse.

DETAILED DESCRIPTION:
In patients medically treated for prosthetic valve infection (PVE), identification of persistent infection or of cure could be very useful to 1/ patients referral to high-risk surgery, 2/ initiation of suppressive antibiotic therapy, or 3/ simplify the follow-up in other patients. The hypothesis is that FDG-PET could thus identify patients at increased risk of recurrence in case of persistent pathological uptake In patients with prosthetic endocarditis and pathological valvular FDG uptake on the initial FDG-PET and not referred to valve replacement at the acute phase, the main objective is to estimate the proportion of those still showing pathological valvular FDG uptake after curative antibiotic treatment. The secondary objectives are 1/ to quantitatively compare the valvular FDG-PET uptake for each individual before and after treatment; 2/ to determine the proportion of those in whom extracardiac foci persist at the end of treatment ; 3/ to evaluate the association between valvular FDG uptake on PET at the end of treatment and PVE relapse at 6 months; 4/ to evaluate the diagnostic performance of an automatic analysis by artificial intelligence of FDG uptake before and after treatment to predict PVE relapse at 6 months.

This is a single-center prospective cohort study. The population is composed of 50 adults with definite PVE according to the ESC 2015 classification, not operated in the acute phase and with pathological FDG-PET at the beginning of curative antibiotic treatment.

A change in practices regarding the duration of antibiotic therapy and the use of valve replacement surgery and its potential complications would benefit patients and reduce the overall cost related to valve prosthesis infection to the healthcare system."

ELIGIBILITY:
"Inclusion criteria:

* Patient aged 18 or over;
* Have a prosthetic valve implanted surgically or by catheter for at least 3 months;
* Presenting a definite IE on a prosthetic valve (ESC definition in force);
* Having benefited from an FDG-PET examination for diagnostic purposes as part of the treatment revealing pathological hyperuptake at the level of the prosthetic valve AND carried out <15 days after the start of antibiotic therapy for infective endocarditis;
* Absence of cardiac surgical intervention performed for the current episode of AE or planned before the end-of-treatment FDG-PET

Exclusion criteria:

* Patient under legal protection, guardianship or curators;
* Pregnancy, breastfeeding;
* Patient not affiliated to a health insurance scheme or not a beneficiary of a social security scheme;
* Simultaneous participation in a study on FDG-PET;
* Absence of informed consent signed by the patient."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Presence of pathological uptake on the prosthetic valve on FDG-PET | at inclusion
  Presence of pathological uptake on the prosthetic valve on FDG-PET performed after the recommended duration of curative antibiotic treatment

SECONDARY OUTCOMES:
Evolution of the FDG uptake intensity on the prosthetic valve by FDG-PET | at inclusion
  by comparing the FDG uptake intensity on the prosthetic valve between initial and at the end of curative antibiotic treatment FDG-PET
Presence of the intensity of extracardiac uptake on the FDG-PET at the end of curative antibiotic treatment in patients presenting with pathological extracardiac uptake on the initial FDG-PET | at inclusion
  by comparing the intensity of extracardiac uptake between FDG-PET initial and at the end of curative antibiotic treatment
Evolution of the intensity of extracardiac uptake on the FDG-PET at the end of curative antibiotic treatment in patients presenting with pathological extracardiac uptake on the initial FDG-PET | at inclusion
  by comparing the intensity of extracardiac uptake between FDG-PET initial and at the end of curative antibiotic treatment
Relapse of endocarditis defined by the same location and the same microorganism within 6 months | 6 month
Therapeutic impact of end-of-treatment PET-FDG measured by stopping or continuing antibiotic treatment | 6 month
  measured by stopping or continuing antibiotic treatment
Diagnostic performance of AI to predict relapse of endocarditis defined by the same location and the same microorganism within 6 months | 6 month
  classification

CONTACTS AND LOCATIONS:
Overall Officials: François Rouzet, MD, PHD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France, France

IPD SHARING:
Plan to Share IPD: Undecided